CLINICAL TRIAL: NCT05564078
Title: A Single-centre, Observational, Prospective Study to Investigate the Effect of IL-13/IL-4 Blockade on Reducing Markers of Airway Autoimmunity in Severe Asthmatics
Brief Title: IL-13 Blockade and Airway Autoimmunity in Asthma
Acronym: IL-SAA
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 14816
Record Dates: First submitted 2022-09-30; First posted 2022-10-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Airway Auto Immunity in Asthma
Keywords: auto immune; severe asthmatics; exacerbations; eosinophilic Asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Subjects with Eosinophilic Asthma
- Subjects without Asthma

SUMMARY:
It has been observed that certain section of patients having severe to moderate Asthma, do not benefit from oral corticosteroids and IL-5 blocking biologics. There is increasing evidence that Airway auto immunity may be responsible for this poor response to treatment. It has been seen in earlier study done at Nair lab that these patients might benefit from Dupilumab, a biologic blocking IL-13/ IL-4. IL-13/IL-4 are the cytokines responsible for increased inflammation in these Asthmatics. The hypothesis is that blocking IL-13/IL-4 will also reduce the airway auto immunity which can be measured by comparing the auto immune markers in airway at baseline (before starting Dupilumab) and 16 weeks (after 4 months of Dupilumab treatment.

DETAILED DESCRIPTION:
Asthma, a chronic airway disease characterized by reversible airflow, airway inflammation and hyper responsiveness. A prominent phenotype is eosinophilic asthma, with a prevalence rate of ~50% and characterised by blood eosinophils >300 cells/μL and sputum eosinophils >3%. Inhaled corticosteroids (ICS) have been successful for treatment of mild-to-moderate asthma. However, ~10% of eosinophilic asthmatics remain uncontrolled despite being on high dose oral corticosteroids. This small percentage contributes disproportionately to 80% of asthma healthcare costs [8-10]. As a steroid-sparing strategy, monoclonal antibody (mAb) therapies targeting interleukin (IL)-5 signalling have been developed that are projected to benefit this difficult-to-treat population. Yet, a subset (30-50%) of them remain symptomatic despite being on oral corticosteroids (OCS) and adjunct anti-IL-5 mAb. Anti- eosinophil peroxidase (EPX) Immunoglobulin G (IgG) levels in the airways strongly correlated with the presence of other auto antibodies, in particular the anti-nuclear antibodies (ANAs) as well as various clinical features of asthma severity. Therefore, a better understanding of the underlying pathology with subsequent identification of clinical/molecular biomarkers remains an unmet clinical need for optimal asthma management. Airway autoimmune responses in severe asthma is an important contributor to airway mucus and this can be ameliorated by blocking the IL-4/IL-13 inflammatory axis.

ELIGIBILITY:
Inclusion Criteria:

* Prior to the beginning of the study, patients must be willing and fully capable to provide written informed consent
* Subjects must be able and willing to comply with the study protocol
* Asthma diagnosed by a respiratory physician ≥ 36 months prior to study enrollment based on the Global Initiative for Asthma (GINA) 2014 guidelines
* Patients referred or routinely followed for asthma by Dr. Nair
* Clinical indication to prescribe dupilumab or will enter a clinical trial where patient will receive drug for at least 4 months
* ICS dose ≥ 500 mcg of fluticasone equivalent/day, and/or daily prednisone

Exclusion Criteria:

* Current smoker defined as having smoked at least one cigarette (or pipe, cigar, or marijuana) per day for ≥ 30 days within the three months prior to screening
* Ex-smokers with ≥ 20 pack-year smoking history
* Current pregnancy or lactation
* Treatment with anti- Immunoglobulin E (IgE), anti-IL-5, or anti-IL-5 Receptor targeted therapy currently or within three months prior to Visit 1
* Any prior medical conditions or treatment history that the physician deems unfit (including but not restricted to chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis).

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severe asthmatics on newly prescribed Dupilimab.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
The proportion of severe asthmatics with a reduction in anti-EPX IgG in airway secretions (marker of airway autoimmunity) | 12 weeks
  Reduction in anti-EPX IgG

SECONDARY OUTCOMES:
To determine the effect of dupilumab on luminal plugging (CT mucus score) and airway obstruction (FEV1) from baseline to post 4 months of therapy | 12 weeks
  CT mucus score
To associate changes with respect to clinical indices of asthma control: blood eosinophils, fractional exhaled nitric oxide (FeNO) and asthma control questionnaire (ACQ) | 12 weeks
  Blood eosinophil count
To determine the changes in sputum composition (sputum eosinophils, neutrophils, free eosinophil granules) and inflammatory mediators (eosinophil peroxidase, T2 cytokines and chemokines) from baseline to post 4 months of therapy | 12 weeks
  Sputum cell differential count

CONTACTS AND LOCATIONS:
Overall Officials: Manali Mukherjee, PHD, Principal Investigator — McMaster University
Locations (1):
- The Research Institute of St. Joe's Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No